CLINICAL TRIAL: NCT04551586
Title: A Phase 1 Study to Assess the Relative Bioavailability of ACH-0145228 When Administered as Immediate Release Tablet Versus Powder-In-Capsule in Healthy Adult Subjects
Brief Title: A Study to Assess ACH-0145228 When Administered as Immediate Release Tablet Versus Powder-In-Capsule in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ACH228-004
Record Dates: First submitted 2020-09-10; First posted 2020-09-16 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-11

CONDITIONS: Healthy
Keywords: Factor D Inhibitor; Complement; Bioavailability; Tablet; Capsule

STUDY DESIGN:
Intervention Model Description: This will be a 3-sequence, 3-period crossover study in healthy adult participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sequence 1 (Experimental): Participants will receive ACH-0145228 once each Period as a single dose under fasted or fed conditions as follows:
  Period 1: ACH-0145228 as an immediate-release tablet under fasted conditions (test-fasted).
  Period 2: ACH-0145228 as an immediate-release tablet under fed conditions (test-fed).
  Period 3: ACH-0145228 as power-in-capsule under fasted conditions (reference).
  There will be a washout period of at least 5 days between each ACH-0145228 dosing.
  Interventions: Drug: ACH-0145228: Immediate Release; Drug: ACH-0145228: Powder-in-capsule
- Sequence 2 (Experimental): Participants will receive ACH-0145228 once each Period as a single dose under fasted or fed conditions as follows:
  Period 1: ACH-0145228 as an immediate-release tablet under fed conditions (test-fed).
  Period 2: ACH-0145228 as power-in-capsule under fasted conditions (reference).
  Period 3: ACH-0145228 as an immediate-release tablet under fasted conditions (test-fasted).
  There will be a washout period of at least 5 days between each ACH-0145228 dosing.
  Interventions: Drug: ACH-0145228: Immediate Release; Drug: ACH-0145228: Powder-in-capsule
- Sequence 3 (Experimental): Participants will receive ACH-0145228 once each Period as a single dose under fasted or fed conditions as follows:
  Period 1: ACH-0145228 as power-in-capsule under fasted conditions (reference).
  Period 2: ACH-0145228 as an immediate-release tablet under fasted conditions (test-fasted).
  Period 3: ACH-0145228 as an immediate-release tablet under fed conditions (test-fed).
  There will be a washout period of at least 5 days between each ACH-0145228 dosing.
  Interventions: Drug: ACH-0145228: Immediate Release; Drug: ACH-0145228: Powder-in-capsule

INTERVENTIONS:
Drug: ACH-0145228: Immediate Release — ACH-0145228 (240 milligrams) will be administered orally on Day 1.
  Other Names: ALXN2050
Drug: ACH-0145228: Powder-in-capsule — ACH-0145228 (240 milligrams) will be administered orally on Day 1.
  Other Names: ALXN2050

SUMMARY:
This will be an open-label, 3-sequence, 3-period crossover study in healthy adult participants to assess the relative bioavailability of ACH-0145228 when administered as an immediate release tablet versus powder-in-capsule.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index in the range of 18.0 to 32.0 kilograms (kg)/meter squared, inclusive, with a minimum body weight of 50.0 kg at screening.
2. No clinically significant history or presence of electrocardiogram findings at screening.
3. Non-sterile male participants must agree to abstinence or use a highly effective method of contraception.
4. Female participants must be of non-childbearing potential and need not employ a method of contraception.

Exclusion Criteria:

1. Clinically significant laboratory abnormalities.
2. History of any medical or psychiatric condition or disease that might limit the participant's ability to complete or participate in this clinical study, confound the results of the study, or pose an additional risk to the participant by their participation in the study.
3. History or presence of drug or alcohol abuse within previous 2 years, current tobacco user, and positive drugs-of-abuse screen and alcohol screen at screening or Day -1 of Period 1.
4. History or presence of clinically significant seizures, head injury, or head trauma.
5. History of procedures that could alter absorption or excretion of orally administered drugs.
6. History of meningococcal infection, or a first-degree relative with a history of meningococcal infection.
7. A history of significant multiple and/or severe allergies or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs.
8. Body temperature ≥ 38.0°Celsius at screening or prior to first dosing in Period 1 or history of febrile illness, or other evidence of infection, within 14 days prior to (first) dosing.
9. Is a female of childbearing potential.
10. Donation of whole blood from 3 months prior to first dosing, or of plasma from 30 days before first dosing, and receipt of blood products within 6 months prior to first dosing.
11. Participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives (if known) or 30 days before first dosing, whichever is longer.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2020-10-19 (Actual)

PRIMARY OUTCOMES:
Relative Bioavailability Of ACH-0145228 Immediate Release Tablet And Powder-In-Capsule | Up to 72 hours postdose
  Relative bioavailability will be measured by the ratio of the area under the concentration versus time curve from time 0 extrapolated to infinity (AUC0-inf).

SECONDARY OUTCOMES:
Area Under The Concentration Versus Time Curve From Time 0 To The Last Measurable Concentration (AUC0-t) Of ACH-0145228 Immediate-release Tablet Under Both Fed And Fasted Conditions | Up to 72 hours postdose
AUC0-inf Of ACH-0145228 Immediate-release Tablet Under Both Fed And Fasted Conditions | Up to 72 hours postdose
Maximum Observed Concentration (Cmax) Of ACH-0145228 Immediate-release Tablet Under Both Fed And Fasted Conditions | Up to 72 hours postdose
Time To Maximum Observed Concentration (Tmax) Of ACH-0145228 Immediate-release Tablet Under Both Fed And Fasted Conditions | Up to 72 hours postdose
AUC0-t Of ACH-0145228 Powder-in-capsule Under Fasted Conditions | Up to 72 hours postdose
AUC0-inf Of ACH-0145228 Powder-in-capsule Under Fasted Conditions | Up to 72 hours postdose
Cmax Of ACH-0145228 Powder-in-capsule Under Fasted Conditions | Up to 72 hours postdose
Tmax Of ACH-0145228 Powder-in-capsule Under Fasted Conditions | Up to 72 hours postdose
Number Of Participants With Treatment-emergent Adverse Events | Day 1 (postdose) through follow-up (30 [+/- 2] days after last study drug administration)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Site, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No